CLINICAL TRIAL: NCT00537745
Title: Vivitrol for Reducing Driving While Impaired Behavior Among Repeat Offenders-a Pilot Study
Brief Title: Vivitrol for Reducing Driving While Impaired Behavior Among Repeat Offenders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pacific Institute for Research and Evaluation (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Principal Investigator, Sandra Lapham, Center Director, Pacific Institute for Research and Evaluation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C18816/6075/DP/US; 0328.01.01
Record Dates: First submitted 2007-09-28; First posted 2007-10-01 (Estimated); Results first posted 2012-08-27 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2012-08

CONDITIONS: Alcohol Consumption
MeSH Terms: conditions — Alcohol Drinking | interventions — vivitrol; Drug Therapy; Medication Therapy Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vivitrol (Experimental): Vivitrol 380 mg/monthly, plus individual compliance enhancement therapy (Medication Management Therapy).
  Interventions: Drug: Vivitrol (Medication Therapy); Other: Medication Management Therapy

INTERVENTIONS:
Drug: Vivitrol (Medication Therapy) — Vivitrol 380 mg/monthly
Other: Medication Management Therapy — Medication Management Therapy once a month.

SUMMARY:
The purpose of this study is to determine whether Vivitrol is effective at reducing attempts to drive after drinking among repeat driving while intoxicated (DWI) offenders with Ignition Interlock devices.

DETAILED DESCRIPTION:
We propose to conduct an open label trial of Vivitrol in combination with an individual compliance enhancement therapy known as Medication Management Therapy (MMT) as an adjunct to Ignition Interlock in the management and treatment of DWI. Subjects will be recruited from a local Interlock provider. This program of research will collect pilot data for a study to determine whether pharmacotherapy, previously recognized as effective, can be successfully combined with existing counseling treatments and sanctions for persons convicted of a repeat DWI alcohol offense. We will investigate the extent to which this combination of sanctions and treatment will significantly decrease attempts to drive after drinking among offenders, and whether the effect persists following discontinuation of Vivitrol.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18
* Capable of understanding and complying with the protocol, and has signed the informed consent document
* Been convicted of a DWI offense, have at least one additional arrest for DWI, and be entering an ignition interlock program
* They must be able to participate in a 6 month outpatient study; and reside within a one-hour commute to the research site
* Women of childbearing potential must have a negative pregnancy test, use contraceptive methods, and not be breastfeeding
* Negative urine toxicological screen for opiates at screening and randomization
* Has a non-custodial stable residence and telephone

Exclusion Criteria

* Is pregnant and/or currently breastfeeding
* Has a clinically significant medical condition or observed abnormality that is contraindicated for Vivitrol treatment
* Is taking an excluded medication, including but not limited to benzodiazepines, anticonvulsants, opiates, or alcohol treatment medication
* Not stable on current anti-depressant, as evidenced by less than 3 months at current dosage, plans to discontinue, or plans to change the dosage
* Has been hospitalized for medical detoxification within 30 days of screening
* Has evidence of severe kidney, heart, or lung disease
* Has evidence of severe hepatic disease (as evidence by BUN > 10% above ULN, AST, ALT > 3x ULN, and GGT > 5x ULN at randomization)
* Known or suspected hypersensitivity to naltrexone and/or Vivitrol in particular
* Current diagnosis and symptoms of major depression, anxiety disorder, mania or psychosis (subjects with their illness in remission for 3 months may be included)
* Opioid use within the past 14 days and/or current or recent (within the past year) diagnosis of dependence or abuse of opiates, benzodiazepines, or cocaine.
* Current or anticipated need for prescribed opiate medication during the study period
* Medication with naltrexone, disulfiram, acamprosate or other medication used to treat alcoholism within the past 30 days
* Impending incarceration or other known situation that would preclude participation in the study
* Other non-alcohol Axis I substance dependence diagnosis in the past 12 months, excluding nicotine, marijuana, and caffeine
* Has participated in a clinical trial of a pharmacological agent within 30 days of screening
* Has any finding that in the view of the principal investigator would compromise the subject's ability to fulfill the protocol visit schedule, and/or visit requirements or would affect subject safety during participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Lapham, MD, MPH, Principal Investigator — Pacific Institute for Research and Evaluation
Locations (1):
- Behavioral Health Research Center of the Southwest, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were initially recruited from only two local Ignition Interlock providers. Recruitment was expanded by placing advertisements in local free press venues and flyers at all local Ignition Interlock providers.
Period: Overall Study
Arm/Group | Vivitrol
Started | 14 (There were three screen fails and two early terminations.)
Began Intervention | 11
Completed | 9
Not Completed | 5
Not completed — Did not meet eligibility criteria | 2
Not completed — Withdrawal by Subject | 2
Not completed — Subject unable to provide Interlock info | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vivitrol
Number analyzed (Participants) | 14
Age Continuous [Mean (Standard Deviation); unit: years] | 43.14 (11.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Average Drinks/day [Mean (Standard Deviation); unit: Standard Drinks] | 3.0 (1.8)
% days w/1+Interlock test failures [Mean (Standard Deviation); unit: percent of days] — The describes the percent of days in the 90 days preceding study screening that the subject had at least 1 interlock test failure.
  percent of days | 3.1 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: Evidence of Attempts to Drive After Drinking
Description: This was measured as Percent of days with an Interlock report of "Failure to Start" due to alcohol pre/on medication and 6 months post medication.
Time Frame: 6 months
Population: Twelve subjects were consented. One was dropped because of no interlock device. Another subject completed Visit 1 and then decided she did not want to receive any injections. Of the ten remaining subjects, seven received all 3, one received 2, and two received only 1, injection. These 10 subjects were used in the intent to treat analysis.
Measure: Mean (Full Range); unit: percent of days
Units Other Than Participants: Percent of Days
Groups:
- Participants: Intervention Group
Arm/Group | Participants
Number analyzed (Participants) | 10
Number analyzed (Percent of Days) | 1000
percent of days
  Percent Days Interlock Fail Pre/on Medication | -1.29 [-6.41 to 2.16]
  Percent Days Interlock Fail Post Medication | -0.30 [-3.23 to 2.13]

2. Primary Outcome: % Days w/1+Interlock Test Failures
Description: This describes the percent of days in past month where the subject at least 1 interlock test failure.
Time Frame: One month post treatment
Population: as for outcome 1
Measure: Mean (Full Range); unit: percent of days
Arm/Group | Vivitrol
Number analyzed (Participants) | 10
percent of days | -.30 [-3.23 to 2.13]

ADVERSE EVENTS:
Arm/Group | Vivitrol
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 1/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Vivitrol (N=12)
Induration at Injection site (Skin and subcutaneous tissue disorders) | 1/10 (1) — Induration at injection site. The area of induration at the injection site gradually subsided and was not palpable at the end of the study.
Nausea (Gastrointestinal disorders) | 1/10 (2)

LIMITATIONS AND CAVEATS:
Fourteen subjects were consented, and began the screening process. Two subjects did not meet entry criteria and 1 withdrew consent prior to injection. Of the remaining 11 subjects, 7 received 3, 2 received 2, and 2 received 1 injection(s).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No